CLINICAL TRIAL: NCT00947726
Title: Ceramide Containing Multivesicular Emulsion Application as a Skin Hydration Treatment for Feet of Subjects With Non-insulin Dependent Diabetes Mellitus.
Brief Title: Ceramide Containing Multivesicular Emulsion Application . . .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Adelaide A. Hebert, MD, The University of Texas Health Science Center at Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK7676 (completed)
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Foot Transepidermal Water Loss in Patients in NIDDM; Foot Dryness in Patients With NIDDM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CeraVe — Using OTC cream on foot twice daily for two weeks.
  Other Names: Ceramide based foot cream

SUMMARY:
We believe that using a ceramide based foot cream two times a day for two weeks will prevent water loss and overall foot dryness in patients with non-insulin dependent diabetes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* non insulin-dependent diabetes
* moderate to severe xerosis of both feet [a score of at least 4 on a scale of 0 (normal) to 8 (deep fissuring)]
* capable of understanding and signing consent form

Exclusion Criteria:

* history of ichthyosis vulgaris
* known hypersensitivity to the topical product used in the study
* previous use of high potency steroids (class I and II) in past 2 week
* presence of acute skin disease or infection, such as vasculitis or cellulitis
* presence of foot ulcer
* evidence of gangrene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Decrease transepidermal water loss and foot dryness in study subjects. | 5 weeks